CLINICAL TRIAL: NCT01116154
Title: A Phase I Study of the Combination of Lenalidomide With the Histone Deacetylase Inhibitor, Vorinostat in Hodgkin and Non Hodgkin's Lymphoma
Brief Title: Vorinostat and Lenalidomide in Treating Patients With Relapsed or Refractory Hodgkin Lymphoma or Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor withdrew support for the study
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Popplewell, Leslie, City of Hope
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08144; NCI-2010-00947 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-04-30; First posted 2010-05-04 (Estimated); Last update posted 2010-12-09 (Estimated); Status verified 2010-12

CONDITIONS: Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Peripheral T-Cell Lymphoma; Post-transplant Lymphoproliferative Disorder; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Testicular Lymphoma; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — Lenalidomide; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive oral vorinostat twice daily on days 1-14 and oral lenalidomide once daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lenalidomide; Drug: vorinostat; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: lenalidomide — Given orally
  Other Names: CC-5013; IMiD-1; Revlimid
Drug: vorinostat — Given orally
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
RATIONALE: Vorinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Biological therapies, such as lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing. Giving vorinostat together with lenalidomide may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of vorinostat when given together with lenalidomide in treating patients with relapsed or refractory Hodgkin lymphoma or non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability of the combination of lenalidomide and vorinostat.

II. To determine the maximum tolerated dose (MTD) and recommended dose of vorinostat and lenalidomide when given in combination in this patient population.

SECONDARY OBJECTIVES:

I. To obtain preliminary data for response rate, time to response, response duration and time to progression (TTP) for vorinostat and lenalidomide when used in combination.

OUTLINE: This is a dose-escalation study of vorinostat.

Patients receive oral vorinostat twice daily on days 1-14 and oral lenalidomide once daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months.

ELIGIBILITY:
Inclusion

* Understand and voluntarily sign an informed consent form
* Able to adhere to the study visit schedule and other protocol requirements
* Patients must have a history of biopsy-documented Hodgkin or non-Hodgkin lymphoma (either B or T cell) and with relapsed or refractory disease after at least one prior line of therapy
* All previous cancer therapy, including radiation, hormonal therapy and surgery, must have been discontinued at least 4 weeks prior to treatment in this study
* Patients must have measurable disease by CT scan; PET scans are desirable but not mandatory, so that patients with negative PET scans but measurable disease by CT are eligible
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 at study entry
* Patients may be enrolled who relapse after autologous stem cell transplant or after allogeneic transplant; they must have no active related infections (i.e., fungal or viral), no acute graft versus host disease (GvHD) of any grade, and no chronic GvHD other than mild skin, or, or ocular GvHD not requiring systemic immunosuppression
* Laboratory test results within these ranges:
* Absolute neutrophil count >= 1,000/mm^3
* Platelet count >= 75,000/mm^3
* Serum creatinine =< 1.5 mg/dL
* Total bilirubin <= 1.5 mg/dL (however, patients with elevation of unconjugated bilirubin alone, as in Gilbert's disease, are eligible)
* AST (SGOT) =< 2 x upper limit of normal (ULN)
* ALT (SGPT) =< 2 x ULN
* Disease free of prior malignancies for >= 5 years with exception of currently treated blast cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* All study participants must be registered into the mandatory RevAssist program and be willing and able to comply with the requirements of RevAssist
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/ml within 10-14 days prior to and again within 24 hours of prescribing lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control-one highly effective method and one additional effective method AT THE SAME TIME-at least 28 days she starts taking lenalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy
* Able to take aspirin or low molecular weight heparin as prophylactic anticoagulation
* Life expectancy greater than 3 months
* Able to swallow enteral medications

Exclusion

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Pregnant or breast-feeding females; lactating females must agree not to breastfeed while taking lenalidomide
* Any condition, including the presence of laboratory abnormalities, that places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Use of any other experimental drug or therapy with 28 days of baseline
* Known sensitivity to thalidomide or histone deacetylating agents
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
* Any prior use of lenalidomide, vorinostat, or other histone deacetylase inhibitors other than valproic acid, which must be stopped 2 weeks prior to study unless being used for seizure control
* Concurrent use of other anti-cancer agents or treatments
* Known positive for HIV or infectious hepatitis type B or C
* Patients with known brain/CNS metastases
* Patients with feeding tubes
* Any history of deep vein thrombosis (DVT) or pulmonary embolism (PE)
* Any current infection requiring the use of antibiotic, antiviral, or antifungal medication
* Any uncontrolled dysrhythmias
* Baseline QTcF interval > 500 msec in the absence of correctable electrolyte imbalance or any patient with a congenital history of QTc prolongation
* Current therapeutic anti-coagulation
* Any contraindication to safely using prophylactic anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Assessment of the Maximum Tolerated Dose and Dose-Limiting Toxicities of the combination of vorinostat and lenalidomide in this patient population | Following Cycle 1 of treatment

SECONDARY OUTCOMES:
Number of patients with Grade 3 or above adverse events | Day 8 and 22 of Cycle 1 and Day 1 of subsequent cycles and Day 30 following the last dose of study drug
Duration, intensity, and time to onset of toxicities | Day 8 and 22 of Cycle 1 and Day 1 of subsequent cycles and Day 30 following the last dose of study drug
AE, laboratory safety assessments, ECOG, ECGs, vital signs, transfusions, hospital days, and antibiotic use | Day 8 and 22 of Cycle 1 and Day 1 of subsequent cycles and Day 30 following the last dose of study drug
Objective response rate | Every nine weeks on therapy after 2 years a minimum of every 6 months
Time to response | Every nine weeks on therapy after 2 years a minimum of every 6 months
Response duration | Every nine weeks on therapy after 2 years a minimum of every 6 months
Progression-free survival | Every nine weeks on therapy after 2 years a minimum of every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Popplewell, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States